CLINICAL TRIAL: NCT00166231
Title: Understanding Pediatric Symptoms and Other Symptoms
Brief Title: Understanding Pediatric Chest Pain and Other Symptoms
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Collaborators: University of Georgia (Other); Children's Healthcare of Atlanta (Other)
Responsible Party: Principal Investigator, Robert Campbell, MD, Professor, Emory University
Other Study IDs: IRB00021881
Record Dates: First submitted 2005-09-13; First posted 2005-09-14 (Estimated); Last update posted 2015-02-25 (Estimated); Status verified 2015-02

CONDITIONS: Chest Pain
Keywords: Innocent heart murmurs; Chest pain; pediatric Cardiology; Somatization; life stress
MeSH Terms: conditions — Chest Pain; Stress, Psychological

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Chest pain patients
- Murmur group

SUMMARY:
The causes of pediatric pain are often not the same for every child. Most children who visit a cardiology specialist with complaints of chest or other somatic pain have no known medical diagnosis to explain their symptoms. These children and their families often leave with no explanation for the child's distress.

This early study will ask parents and children specific questions related to the stress in their lives, their emotional well-being and the children's physical functioning. The investigators want children who experience chest and other somatic pain, and those who do not, to be in their study so that they can look at both groups.

The investigators hope to use these answers to better inform cardiologists who often work with children with non-cardiac pain and, in turn, help them to better serve their patients. Ultimately, the investigators hope that the answers they get will provide answers to these families. They also hope to use the results of this study to put together a short screener for the cardiologist to give to pediatric patients with complaints of chest or other somatic pain to help the cardiologists better understand their patients' symptoms.

DETAILED DESCRIPTION:
The current investigation will address some similar factors considered in prior research, but will considerably extend our understanding of how psychological, familial, and environmental factors influence noncardiac chest pain. In this investigation, a number of variables that have not been considered in prior research in this area will be included. Among these child variables are: the children's pain coping strategies, the children's somatization behaviors aside from chest pain, the children's externalizing symptoms (e.g., symptoms of ADHD, oppositional defiant disorder), school related problems, social competencies, parental perceptions of the child's vulnerability, functional disability (the degree to which chest pain interferes with normal daily functioning), and the child's health care utilization. Also, a more sensitive quantification of the children's frequency and intensity of chest pain will be collected, as well as information on situations in which the pain occurs. Parent report of child functioning and child self-report will be used to assess children's behavior. The parental factors to be assessed include the parents' own physical conditions and health care utilization, as well as the parents' psychological functioning. The amount of changes and stress the family as a whole has experienced in different domains will also be assessed as well. Measures of these constructs, as well as children's anxiety and depression (similar to Lipsitz et al. reviewed above) will be collected at the time of the original appointment.

With the exception of the chest pain measure, quantification of these variables will be collected for both chest pain and innocent murmur patients between the ages of 8 and 18 years of age at the time of their initial appointment. Further, approximately one month following the medical assessment by the cardiologists, the parents and children will be asked to complete a measure of their satisfaction with the medical care they were provided, their health care utilization subsequent to the diagnostic cardiology appointment, their various somatic symptoms, and their functional disability at the one month follow-up assessment. Also, the chest pain patients will be asked to complete the chest pain inventory in conjunction with their parent.

Between-group analyses will address how these multiple variables differ for the chest pain group and patients presenting for an evaluation for heart murmurs. This will be true at both the time of the patients' appointment and at follow-up. Further, within-group correlational analyses will be conducted primarily for with the chest pain group. The goal of these within group analyses will be to address how the various child, parent, and familial factors correlate with the children's chest pain symptoms, healthcare utilization, other somatic symptoms, and functional disability. In addition, for the chest pain group, the patients' and their families' functioning at the time of the initial appointment will be used to predict chest pain and other somatic symptom maintenance, health care utilization following the initial appointment, and satisfaction with their medical care at follow-up. Each of these questions will advance the literature in this area.

We should also point out why the innocent murmur group was chosen as a comparison sample for the chest pain patients. As noted above, pain is a subjective experience that is first noted by the patient and then communicated to others. It is then reacted to in various ways by those in the child's environment. In contrast, a child with a heart murmur is not the one who first notices the symptom and then communicates it. Instead, the patient with a murmur is told that they have the symptom by a pediatrician, family practice physician, or other health care provider. This tendency to notice and interpret pain in a particular manner is an essential component in the history of the children and their families who report to cardiology clinics for an evaluation of the etiology of chest pain. Such noticing and interpretation is fundamentally a psychological process.

Comparison: adolescents who present in a cardiac specialty clinic with noncardiac chest pain versus those who present with innocent murmurs.

ELIGIBILITY:
Inclusion Criteria:

* 8-18 years of age
* Pediatric patients with referrals for innocent heart murmurs
* Pediatric patients experiencing chest pain
* English speaking

Exclusion Criteria:

* Non English speaking patients

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: enrolling pediatric patients with either chest pain or innocent heart murmur referrals
Sampling Method: Non-Probability Sample
Enrollment: 156 (Actual)
Dates: Start 2004-03; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Change in Children Depression Inventory | Baseline, 4 weeks
  Children Depression Inventory (CDI) is a 27-item self-report scale of depressive symptoms suitable for use by youth ranging from 7 to 17 years. The 27 items on the assessment are grouped into five major factor areas. The item score are rated 0-2 with a total scores summed and converted to T scores. The total T score ranges from 33 to 100 with high scores indicating higher levels of depressive symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Robert M Campbell, MD, Principal Investigator — Emory University; Ronald L. Blount, PhD, Principal Investigator — University of Georgia; Greg Johnson, MD, Principal Investigator — Emory University; Rose Cummings, DO, Principal Investigator — Emory University; Patty Simpson, MSN, Principal Investigator — Emory University; Kenneth Dooley, MD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Childrens Healthcare of Atlanta at Egleston, Atlanta, Georgia
  - Sibley Heart Center Cardiology, Atlanta, Georgia

REFERENCES:
- [Background] Blount RL, Morris JA, Cheng PS, Campbell RM, Brown RT. Parent and child psychological factors in pediatric syncope and other somatic symptoms. J Consult Clin Psychol. 2004 Aug;72(4):597-604. doi: 10.1037/0022-006X.72.4.597. PMID 15301644
- [Background] Claar RL, Walker LS, Smith CA. Functional disability in adolescents and young adults with symptoms of irritable bowel syndrome: the role of academic, social, and athletic competence. J Pediatr Psychol. 1999 Jun;24(3):271-80. doi: 10.1093/jpepsy/24.3.271. PMID 10379142
- [Background] Cohen LL, Blount RL, Cohen RJ, Schaen ER, Zaff JF. Comparative study of distraction versus topical anesthesia for pediatric pain management during immunizations. Health Psychol. 1999 Nov;18(6):591-8. doi: 10.1037//0278-6133.18.6.591. PMID 10619532
- [Background] Massin MM, Bourguignont A, Coremans C, Comte L, Lepage P, Gerard P. Chest pain in pediatric patients presenting to an emergency department or to a cardiac clinic. Clin Pediatr (Phila). 2004 Apr;43(3):231-8. doi: 10.1177/000992280404300304. PMID 15094947
- [Background] Lam JC, Tobias JD. Follow-up survey of children and adolescents with chest pain. South Med J. 2001 Sep;94(9):921-4. PMID 11592755